CLINICAL TRIAL: NCT01900847
Title: Ketamine and Morphine Versus Morphine Alone for the Treatment of Acute Pain in the Emergency Department
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: concern of side effects
Sponsor: University of Arizona (Other)
Collaborators: American College of Emergency Physicians (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-0045
Record Dates: First submitted 2013-07-08; First posted 2013-07-17 (Estimated); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Acute Pain
Keywords: Ketamine; Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Ketamine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine and placebo (Active Comparator): Patient's will receive morphine during the usual course of their emergency department care and will receive a saline in a volume equivalent to the ketamine administered in the experimental arm of the stuy
  Interventions: Drug: Morphine; Drug: placebo
- Morphine and Ketamine (Experimental): Patient's will receive a 0.3mg/kg dose of ketamine in addition to morphine given in the usual course of emergency department care
  Interventions: Drug: Ketamine; Drug: Morphine

INTERVENTIONS:
Drug: Ketamine — 0.3mg/kg ketamine
  Arms: Morphine and Ketamine
Drug: Morphine — Dosage of morphine determined by treating physician
Drug: placebo — saline of same volume as appropriate weight based dose of ketamine
  Arms: Morphine and placebo

SUMMARY:
Our goal is to study whether giving people low dose ketamine along with morphine when they come to the Emergency Department will help their pain more than giving morphine by itself. There have been many studies showing that low dose ketamine is safe and effective for pain control. Ketamine is frequently used for pain control in ambulances and helicopters transporting injured patients to the hospital and has also been used for pain control in people who have just had surgery. The investigators would like to see if low dose ketamine would be safe and effective for patients with pain in the Emergency Department.

Patients are eligible for the study if they come to the Emergency Department and their treating physician decides to treat them with morphine (with certain exceptions such as pregnant patients and patients with eye injuries). They will be given information about participating in the study and if they agree, they will be given the study drug. The study drug will be either ketamine or salt water (saline). If patients continue to be in pain they will continue to receive doses of morphine just as they would if they were not in the study. If the treating physician feels that morphine alone is not enough, they will be free to choose another pain medication as they would normally.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to Emergency Department in acute pain
* age 18 and over
* determined to require morphine for pain control by treating physician

Exclusion Criteria:

* Patients presenting with headache or head injury
* Patient with eye injury or eye pain
* Nontraumatic chest Pain
* Pregnant patients or women of childbearing potential
* Patients allergic to morphine or ketamine
* Patients with known history of narcotic/alcohol abuse or presenting for narcotic medication refill
* Patients with hypertension: diastolic blood pressure > 100 OR systolic blood pressure > 180
* Patient whose pain is so severe that they are unable to give informed consent
* Patients who have had bad experiences to prior hallucinations from any origin

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona Health Network University Campus 1501 North Campbell Ave, Tucson, Arizona, United States

REFERENCES:
- [Background] Berkman, M. R., Larsen, J., Smith, J., Caldwell, J., Waterbrook, A., Stolz, U., & Denninghoff, K. (2014). 369 Ketamine and Morphine versus Morphine Alone for Treatment of Acute Pain in the Emergency Department. Annals of Emergency Medicine, 64(4), S131-S132.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Morphine and Placebo | Morphine and Ketamine
Started | 10 | 7
Completed | 10 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine and Placebo | Morphine and Ketamine | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Customized [Number; unit: participants]
  > 18 years | 10 | 7 | 17
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Females and males | 10 | 7 | 17
Region of Enrollment [Number; unit: participants]
  United States | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Score
Description: Pain 0-10 with 0 being no pain and 10 being the worst pain
Time Frame: Baseline (zero minutes), 30 minutes and 1 hour after receiving study drug
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Morphine and Placebo | Morphine and Ketamine
Number analyzed (Participants) | 10 | 7
score on a scale
  time 0 | 6.9 (2.9) | 7.3 (1.4)
  30 min | 7.7 (2.0) | 3.7 (2.8)
  60 min | 6.8 (1.6) | 4.9 (2.7)

2. Secondary Outcome: Total Amount of Morphine and Other Pain Medications Administered
Time Frame: Data collected from the duration of the patient's Emergency Department stay (expected average 5 hours)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Morphine and Placebo | Morphine and Ketamine
Number analyzed (Participants) | 10 | 7
mg | 9 (5.3) | 10.3 (5.9)

3. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Data collected from the duration of the patient's Emergency Department stay (expected average 5 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine and Placebo | Morphine and Ketamine
Number analyzed (Participants) | 10 | 7
Participants | 4 | 4

ADVERSE EVENTS:
Arm/Group | Morphine and Placebo | Morphine and Ketamine
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 4/10 | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Morphine and Placebo (N=10) | Morphine and Ketamine (N=7)
severe dysphoric reaction (Psychiatric disorders) | 0 | 1
adverse event not specified (General disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No